CLINICAL TRIAL: NCT02814552
Title: OPTImizing Precision of Hypertension Care to Maximize Blood Pressure Control Pilot (OPTI-BP Pilot)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: OneFlorida Clinical Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: IRB201501060
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: High Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Blood Pressure Consented (Other): Participants will have the following performed: medical history and blood pressure levels will be collected, and blood samples. Then using the HTN PRA App recommendation regarding standard of care medication dosing will be adjusted for optimal blood pressure control.
  Interventions: Other: HTN PRA App; Other: Blood Sample
- De-identified historical data (No Intervention): De-identified historical data will be collect based on age (no dates), blood pressure of treated (noted with medications), blood pressure of non-treated (noted without medications), and list of medications. The data will be compared to the High Blood Pressure Consented group to determine the effect of using the HTN PRA App.

INTERVENTIONS:
Other: HTN PRA App — The HTN PRA App will be used to adjust standard of care medication dosages for high blood pressure drugs which may include: thiazide diuretic (water pill), usually called hydrochlorothiazide (HCTZ) or chlorthalidone, and an ACE inhibitor or an angiotensin receptor blocker.
  Other Names: on-line app
  Arms: High Blood Pressure Consented
Other: Blood Sample — Blood sample for plasma renin activity activity will be obtained at least once (at baseline) and if BP is not controlled after 1-3 months, an additional blood sample may be obtained.
  Arms: High Blood Pressure Consented

SUMMARY:
Hypertension (HTN) is a major risk factor for coronary heart disease (CHD), heart failure, kidney failure and stroke. Disparities in HTN prevalence, treatment and control in the US have persisted for decades. The prevalence of HTN is 44% among Blacks, which is among the highest rates in the world. Those in ethnic/racial, rural, socioeconomically disadvantaged and other medically underserved populations are known to have the worst blood pressure (BP) control. Awareness of, treatment for, and control of HTN is not optimal, and varies according to race, whereby BP is controlled in ~53% of non-Latino Whites, 42% of non-Latino Blacks and only 34% of Latinos. Fundamental underlying differences in the pathophysiology contribute to HTN among different race groups. The United States (US) 2014 HTN recommendations outline race-based pharmacotherapy care for HTN. However, these recommendations use race-based population assumptions for Whites and Blacks only, do not include Latino ethnicity and have no accompanying guidelines or tools for successful implementation, particularly in rural primary care practices where disparate populations are common. Moreover, these recommendations only apply to initial therapy and lack guidance on subsequent regimen selection. The Optimizing Precision of HTN Care to Maximize BP Control Pilot (OPTI-BP Pilot), will directly address a long known and growing health disparity concern in the US which includes higher rates of death from CHD and stroke among Blacks and the poorest rates of HTN control among Latinos. Utilizing a mixed methods approach, the overarching goal of OPTI-BP Pilot is to test, using a pragmatic trial design, a personalized, algorithmic-based HTN management approach focused on age, race, biomarker (plasma renin activity) and treatment factors. The investigators hypothesize that implementation of a precision-based approach to the care of HTN in the community will improve BP reduction and ultimately reduce risk for CHD, stroke and death among those most affected by HTN.OPTI-BP Pilot is significant because it will utilize an innovative, systematic, precision-focused HTN management approach in an underserved, diverse population where BP control is currently suboptimal and lays the infrastructure groundwork for broad implementation across all areas of the US to minimize HTN related disparities and improve HTN outcomes.

DETAILED DESCRIPTION:
The purpose of this research study is to develop pilot data to support a more precise way to treat high blood pressure based on an individual person's specific characteristics. Information from a blood test called plasma renin activity will be entered into an on-line app that may more precisely determine which medication should be used to treat high blood pressure than random selection. Renin is a substance in the body that is known to affect your blood pressure. By measuring plasma renin activity, and using that to select a blood pressure lowering medication it may help to more precisely select medications based on how an individual will respond.

ELIGIBILITY:
Inclusion Criteria:

* untreated HTN (systolic BP ≥ 140 or diastolic BP ≥ 90 mm Hg while taking no anti-HTN drugs)
* treated, uncontrolled HTN (systolic BP ≥ 140 or diastolic BP ≥ 90 mm Hg while taking one or more anti-HTN drug)
* provide voluntary, written informed consent
* willing to comply with requirements of the study including provision of a blood sample for local laboratory determined PRA.

Exclusion Criteria:

* treated and controlled HTN (systolic BP < 140 mm Hg and diastolic BP < 90 mm Hg)
* systolic BP ≥ 180 mm Hg or diastolic BP ≥ 110 mm Hg
* secondary forms of HTN or any active, unstable disease process requiring new diagnostic and therapeutic plans
* any life-threatening illness
* history of alcohol or drug abuse in the past 5 years
* mental illness or personality disorder that might interfere with adherence to study protocol
* end-stage renal disease and progressive chronic kidney disease with serum creatinine >2.5 mg/dl
* intolerance to two or more classes of anti-HTN medications
* pregnant women or breast feeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-06-18 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
BP control | 6 months
  We will measure BP control in patients who underwent PRA testing. BP control in the PRA tested patients will be compared with historic control patients who did not undergo PRA testing.

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda M Cooper-DeHoff, PharmD, MS, Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - UF Health Family Medicine, Macclenny, Florida
  - UF Health Family Medicine - Old Town, Old Town, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mehanna M, Chen YE, Gong Y, Handberg E, Roth B, De Leon J, Smith SM, Harrell JG, Cooper-DeHoff RM. Optimizing Precision of Hypertension Care to Maximize Blood Pressure Control: A Pilot Study Utilizing a Smartphone App to Incorporate Plasma Renin Activity Testing. Clin Transl Sci. 2021 Mar;14(2):617-624. doi: 10.1111/cts.12922. Epub 2020 Nov 30. PMID 33142006